CLINICAL TRIAL: NCT02101658
Title: Evaluating Expectancy Effects in Weight Loss Measurement
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Gareth R. Dutton PhD, Associate Professor of Medicine, University of Alabama at Birmingham
Other Study IDs: UAB-NORC-expectancy pilot
Record Dates: First submitted 2014-03-26; First posted 2014-04-02 (Estimated); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Accuracy of Clinic-based Weight Measurements

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- weight data assessors: students recruited to weigh individuals in a research-based clinic
  Interventions: Other: clinic-based weight measurements

INTERVENTIONS:
Other: clinic-based weight measurements

SUMMARY:
The purpose of this project is to examine potential bias or expectancies in individuals' measurement and recording of weight in a clinical-research setting.

ELIGIBILITY:
Inclusion Criteria:

* 19+ years-old
* available to attend clinic sessions on dates provided for data collection

Exclusion Criteria:

* younger than 19 years
* not available on specified dates of data collection

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: undergraduate students
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2014-03; Primary Completion 2014-04 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
accuracy of clinic-based weight measurement | baseline
  Participants will be asked to weigh individuals who they have been told are completing either the treatment or control condition of a weight loss trial (individuals will actually be paid actors playing the role of a study participant). Participants will weigh individuals on calibrated balance-beam scales, and the discrepancy between weights recorded when individuals are thought to be a treatment or control participant will be calculated, which is the primary outcome for this study.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States